CLINICAL TRIAL: NCT01550926
Title: A Study to Assess the Pharmacologic Equivalence of Two Orlistat Dosage Forms
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: W3680604
Record Dates: First submitted 2011-11-17; First posted 2012-03-12 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2012-04

CONDITIONS: Overweight
Keywords: orlistat; overweight; bioequivalence
MeSH Terms: conditions — Overweight | interventions — Orlistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Active Comparator): 60 mg orlistat
  Interventions: Drug: 60 mg orlistat
- Arm 2 (Active Comparator): 120 mg orlistat (2 X 60 mg capsules)
  Interventions: Drug: 120 mg orlistat
- Arm 3 (Experimental): orlistat experimental formulation
  Interventions: Drug: orlistat experimental dose

INTERVENTIONS:
Drug: 120 mg orlistat — 2 X60 mg capsule
  Arms: Arm 2
Drug: 60 mg orlistat — 60 mg orlistat
  Arms: Arm 1
Drug: orlistat experimental dose — experimental
  Arms: Arm 3

SUMMARY:
The purpose of this study is to determine whether a new dosage form and dose of orlistat is equivalent to the currently marketed form.

ELIGIBILITY:
Inclusion Criteria:

* age: 18-60 years
* Body Mass Index: 25-33

Exclusion Criteria:

* gastrointestinal disease
* organ transplant
* HIV, hepatitis B or C
* food allergies
* alcohol or other substance abuse
* smoking

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2009-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Fecal fat excretion | 9 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- MDS Pharma Services, Belfast, Northern Ireland, United Kingdom